CLINICAL TRIAL: NCT06073717
Title: Motor-cognitive Training Effects on Cancer-related Cognitive Impairment and Muscle-brain Crosstalk Biomarkers in Breast Cancer Survivors: the BRAINonFIT Study
Brief Title: Motor-cognitive Training Effects on Cognition in Breast Cancer Survivors: the BRAINonFIT Study (BRAINonFIT).
Acronym: BRAINonFIT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Jesus Orellana Jaen, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0570-N-23
Record Dates: First submitted 2023-09-22; First posted 2023-10-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Survivors; Cognitive Impairment; Executive Dysfunction
Keywords: Cancer-related Cognitive Impairment; Physical exercise; dual motor-cognitive tasks; cognitive stimulation; Neurocognitive disorders
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity; Neurocognitive Disorders | interventions — Exercise; Health

STUDY DESIGN:
Intervention Model Description: This study has been designed as a randomised, controlled, longitudinal (20 weeks), three-arm, parallel study with a follow-up phase (12 weeks).
Who Masked: Participant
Masking Description: Regarding the control of experimental bias, simple blinding will be used. Thus, participants will be blinded to the research problem. They will be informed that three interventions will be applied (without comment on specific details of each one) randomly allocated, to compare the impact on cognitive functions, circulating levels of certain biomarkers, and different symptoms associated with breast cancer. Therefore, study participants will not be able to know to which experimental or control group they belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise Intervention (Experimental): This arm will receive a 5-month (20 weeks) supervised exercise program based on aerobic and resistance/strength training together with a weekly calorie or step challenge.
  Interventions: Behavioral: Exercise
- Dual Motor-Cognitive Intervention (Experimental): This arm will receive a 5-month (20 weeks) supervised and simultaneous dual-task program based on aerobic, resistance, and cognitive stimulation training together with a weekly calorie or step challenge
  Interventions: Behavioral: Motor-cognitive Training
- Health and Wellness Intervention (Active Comparator): This arm will receive a 5-month health and wellness program.
  Interventions: Behavioral: Health and Wellness

INTERVENTIONS:
Behavioral: Exercise — Participants will complete a 5-month exercise program structured in 4 blocks of 5 weeks. Three supervised and combined aerobic/strength exercise sessions each week will be performed together with an aerobic weekly challenge. Aerobic exercise will be performed for 20-30 minutes using a treadmill, bicycle, or circuit training at light to moderate intensities (40-75% of heart rate reserve) during the first two blocks; gradually achieving high intensity (>75% of HHR) in the last two blocks. Heart rate and the subjective perception of the exertion scale (6-20 Borg scale) will be monitored. Strength exercises will be started at light to moderate intensities (2 sets of 15-20 repetitions at 40-50% of repetition maximum), performed muscle actions at high intensities in the last two blocks (2 sets of 8-15 repetitions at 50-75% RM); using elastic bands, free weights, and weights gym exercises.
  Arms: Exercise Intervention
Behavioral: Motor-cognitive Training — Participants will complete the same four-block exercise program in terms of type, frequency, intensity, and volume of physical/motor training. Simultaneous with the progression of physical/motor training, the complexity of cognitive stimulation will be increased according to the performance of the participants. General dual-task training will be performed, which describes the use of a physical/motor intervention with different cognitive stimulations (memory, language, intelligence, attention, processing speed, calculation, inhibitory control) that are not specific to the methods to be used for their assessment.
  Arms: Dual Motor-Cognitive Intervention
Behavioral: Health and Wellness — Participants randomly assigned to the health and wellness group will be advised and re-educated to support and improve health aspects. Participants in this group will aim to achieve the physical activity recommendations, and in addition, they will receive bi-weekly emails and phone call coaching with tools to empower patients with knowledge about physical exercise, nutrition, and brain health guidelines. Following completion of the 5-month exercise program, this group will receive an exercise program for 12 weeks.
  Arms: Health and Wellness Intervention

SUMMARY:
The goal of this interventional study is to assess the effects of either physical exercise program or combined with cognitive training (dual motor and cognitive training program) on breast cancer survivors. The main questions it aims to answer are:

* Analyze the effectiveness of a supervised dual-task training program or a physical exercise program on the executive functions of the participants.
* Evaluate the impact of both interventions on physical function, emotional aspects, and important biomarkers related to muscle-brain crosstalk.

Participants will perform a 20-week supervised and controlled program, three times a week, along with weekly calorie and step challenges.

Researchers will compare the dual-task training group, with the physical exercise group, and with a control group, which will perform the guideline recommendations of physical activity (non-supervised) to see how these intervention approaches can impact cognitive functions, physical functions, emotional aspects, and biomarkers related to muscle-brain crosstalk.

Assessments will take place at three-time points: at baseline, after the intervention (20 weeks post-baseline) and after a 12-week follow-up period (32 weeks post-baseline).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage I-IIIA breast cancer
* Completed primary treatment, including surgery, radiotherapy and/or chemotherapy
* Scheduled to receive adjuvant endocrine therapy, or currently receiving adjuvant endocrine therapy
* Without functional limitations or other illnesses that condition and prevent them from practising intense physical exercise
* FACT-Cog questionnaire score ≥ 10th percentile considering age groups
* Fluency in Spanish (spoken and written)

Exclusion Criteria:

* Undergoing radiotherapy and/or chemotherapy
* FACT-Cog questionnaire score ≤ 10th percentile considering age groups
* Congenital heart disease
* Chronic lung disease
* Severe psychiatric disorders
* History of substance abuse, or dependence (other than tobacco)
* Mood disorders require treatment (anxiety or depression)
* Relapses (2-3 months before the study start)

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Executive Function (Cognitive Flexibility and Processing Speed) | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Trail Making Test A and B (minimum and maximum values, defined by the time in seconds, depend on the age- and education-normalised groups; higher scores mean worse results)

SECONDARY OUTCOMES:
Inhibitory Control and Concentration | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Stroop Color and Word test (minimum and maximum values, defined by the time in seconds, depend on the age- and education-normalised groups; higher scores mean worse results)
Verbal Intelligence, Non-verbal Intelligence, Verbal memory, and Non-verbal Memory | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Reynolds Intellectual Assessment Scale (Global index values range from ≤ 69 to ≥ 130, mean value of 100; higher scores mean better results)
Learning Ability | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Wechsler Memory Scale subtest "word pairs" (The subtest score range from 40 to 60, mean value of 100; higher scores mean better results)
Perceived Cognitive Functions | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Functional Assessment of Cancer Therapy: Cognition (FACT-Cog) (Total score ranges from 0 to 148; higher scores mean better results)
Max. Oxygen Consumption | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Modified Bruce Test (80% sub-max)
Muscular Strength of shoulder and knee extensors | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Isokinetic dynamometer
Range of Movement | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Manual Goniometer
Forced Vital Capacity (FVC) and Forced Expiratory Volume (FEV) | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Spirometry (FEV/FVC ratio, represented in percentages)
Volume of physical activity | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Accelerometer (Volume in minutes per week)
Intensity of Physical Activity | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Accelerometer (Intensity in metabolic equivalents)
Weight and Height | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Body Mass Index (weight and height will be combined to report BMI in kg/m^2)
Brain-Derived Neurotrophic Factor (BDNF), Vascular Endothelial Growth Factor (VEGF), Fibroblast Growth Factor 17 (FDF-17), Soluble Klotho (S-KL) | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Concentration of these proteins in plasma by ELISA kit (Concentration of these proteins will be expressed in pg/mL or ng/mL)
Fatigue | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Functional Assessment of Chronic Illness Therapy: Fatigue (FACIT-F) (Total score range from 0 to 52; higher scores mean better results)
Pain Scale | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Visual Analogue Scale (Total score ranges from 0 to 10; higher scores mean worse results)
Depression | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  Back Depression Inventory (Total score ranges from 0 to 63; higher scores mean worse results)
Anxiety | Baseline (week 0); Post-intervention (25 weeks post-baseline); and Post-follow up (32 weeks post-baseline)
  State-Trait Anxiety Inventory (The score ranges from 20 to 80; higher scores mean worse results)

CONTACTS AND LOCATIONS:
Overall Officials: Matilde Mora Fernández, PhD, Study Director — University of Seville; Luis Carrasco Páez, PhD, Study Director — University of Seville; Jesús Orellana Jaén, Principal Investigator — University of Seville
Locations (3):
- Spain (3):
  - SADUS - Servicio de Actividades Deportivas de la Universidad de Sevilla, Seville, Sevilla
  - Laboratorio de Ciencias del Deporte, Seville, Sevilla
  - Oncoavanze, Seville, Sevilla

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jesus OJ, Luis CP, Matilde MF. Effects of exercise on cancer-related cognitive impairment in breast cancer survivors: a scoping review. Breast Cancer. 2023 Nov;30(6):885-909. doi: 10.1007/s12282-023-01484-z. Epub 2023 Jul 22. PMID 37480454
- [Derived] Orellana-Jaen J, Mora-Fernandez M, Carrasco-Paez L. Effects of a motor and cognitive training program on executive function and different biomarkers related to muscle-brain crosstalk in breast cancer survivors: 3-arm randomised controlled BRAINonFIT study protocol. Contemp Clin Trials. 2024 Nov;146:107672. doi: 10.1016/j.cct.2024.107672. Epub 2024 Sep 10. PMID 39265784